CLINICAL TRIAL: NCT01795235
Title: Glucagon, Ghrelin and Growth Hormone as Counterregulatory Hormones
Brief Title: Study of Glucagon, Ghrelin and Growth Hormone as Counterregulatory Hormones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Michael Thorner, MD, MD, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16391
Record Dates: First submitted 2013-02-12; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Sodium Chloride; Glucagon; Injections; Atenolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline s.c. injection and placebo tablet (Other): Saline s.c. injection and one placebo tablet (preceded by one placebo tablet per day at 0900h for two days before admission).
  Interventions: Drug: Saline; Drug: Placebo
- glucagon s.c. injection and placebo tablet (Other): 1 mg glucagon s.c. injection and one placebo tablet (preceded by one placebo tablet per day at 0900h for two days before admission).
  Interventions: Drug: Glucagon; Drug: Placebo
- Saline s.c. injection and atenolol tablet (Other): Saline s.c. injection and 100 mg atenolol tablet
  Interventions: Drug: Saline; Drug: Atenolol
- glucagon s.c. injection and atenolol tablet (Other): 1 mg glucagon s.c. injection and 100 mg atenolol tablet
  Interventions: Drug: Glucagon; Drug: Atenolol

INTERVENTIONS:
Drug: Saline — Saline s.c.
  Other Names: NormalSaline; 0.9% Sodium Chloride Solution
  Arms: Saline s.c. injection and atenolol tablet; Saline s.c. injection and placebo tablet
Drug: Glucagon — Glucagon s.c.
  Other Names: Glucagon for injection
  Arms: glucagon s.c. injection and atenolol tablet; glucagon s.c. injection and placebo tablet
Drug: Placebo — Sugar Pill
  Arms: Saline s.c. injection and placebo tablet; glucagon s.c. injection and placebo tablet
Drug: Atenolol — Beta-1 receptor antagonist
  Other Names: Tenormin
  Arms: Saline s.c. injection and atenolol tablet; glucagon s.c. injection and atenolol tablet

SUMMARY:
Glucagon has been used for decades as a test of growth hormone (GH) reserve. The pathway by which GH is stimulated by glucagon is not established. Acyl ghrelin has been shown to increase GH levels and to be stimulated by an increase in adrenergic activity. The proposed study will test the concept that with the fall in blood glucose it is likely that there is a sympathetic discharge which contributes to the increase in acyl ghrelin and indirectly leads to the increase in GH and cortisol.

DETAILED DESCRIPTION:
Glucagon given to healthy adults in doses of 1-1.5 mg i.m. has been shown to result in a peak glucagon level in the circulation after 30 min, followed by an increase in glucose and insulin levels. The subsequent decline in glucose, insulin and glucagon was followed by an increase in cortisol and GH. Ghrelin is a 28 amino acid peptide which is released from the fundus of the stomach, within the oxyntic glands and the small intestine. It circulates in two major forms, acylated and des-acylated ghrelin. Acylated ghrelin has strong GH-releasing effects which are mediated via the G-protein coupled ghrelin receptor. The proposed study will test the concept that with the fall in blood glucose during a glucagon test it is likely that there is a sympathetic discharge which contributes to the increase in acyl ghrelin and indirectly leads to the increase in GH and cortisol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy normal men
2. Age 18-30 yrs
3. BMI 18-27 kg/m2

Exclusion Criteria:

1. Medication or previous surgery known to affect ghrelin secretion.
2. Medications known to have an impact on body weight (Seroquel, tricyclic antidepressants).
3. Medications known to have an impact on the beta adrenergic system.
4. Coronary artery disease, congestive heart failure, peripheral vascular disease, diabetes mellitus, significant hypertension (BP >180 systolic or >100 diastolic at rest); renal, hepatic, pulmonary disease; untreated hypothyroidism, untreated hyperthyroidism; history of seizure disorder; history of malignancy (other than some skin cancers), history of active chronic infections (e.g., HIV, tuberculosis).
5. Endocrine disorders, i.e., pheochromocytoma, adrenal insufficiency
6. Hematocrit < 41% men
7. History of daily tobacco use within past 3 months
8. Chronic alcohol abuse by history
9. Weight not stable (more than 10% weight change or more over past 6 months)
10. Strenuous exercise for average of more than 60 min/day
11. Investigational drug within past 6 weeks
12. Psychiatric history especially eating disorders
13. Transmeridian travel within 2 weeks prior to or during study
14. Known hypersensitivity to beta-blockers
15. Estimated Glomerular Filtration Rate below 60 mL/min/1.73m2.
16. Known cardiac dysrhythmia, especially first degree heart block. -

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Circulating acyl-ghrelin concentration after glucagon stimulation with and without beta-adrenergic blockade | 18 months

SECONDARY OUTCOMES:
Association between circulating acyl-ghrelin concentration and GH and cortisol after glucagon administration with and without beta-adrenergic blockade | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael O Thorner, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States